CLINICAL TRIAL: NCT01404624
Title: Increased Density of Ghrelin-Expressing Cells in the Gastric Fundus and Body in Prader-Willi Syndrome
Brief Title: Characterization of Transcriptional Regulators of Ghrelin Hormone Which Causes Genetic Obesity
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Dong-Kyu Jin, Samsung Medical Center
Other Study IDs: 2007-01-016
Record Dates: First submitted 2011-07-26; First posted 2011-07-28 (Estimated); Last update posted 2011-07-28 (Estimated); Status verified 2011-07

CONDITIONS: Prader Willi Syndrome; Obesity
MeSH Terms: conditions — Prader-Willi Syndrome; Obesity

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The problem point of the Prader-Willi Syndrome (PWS) patient is the obesity which is intense and the plasma ghrelin level which increases unusual from the recently PWS patients was discovered. The Ghrelin is endogeneous ligand of growth hormone secretagogue receptor with peptide hormone and the location is 3p26-p25. Becomes the secretion even from nervous system but from dignity X/A cell it is secreted mainly and growth is important even in the vagal control against food and intake and a dignity function even on the action outside which promotes the secretion which drives it operates. It increases food intake specially and in order to accomplish the action which diminishes fat utilization the obesity with the week cause which it does the mortar it is thought. Active the ghrelin of the form is essential in hormonal activity of the ghrelin and appetite and growth hormone it participates to the secretion promotion which drives. Action of the Ghrelin measuring the quantitative change in middle acylated of the PWS patient ghrelin in order to happen after the acylation initially by one interest ghrelin which is attempted the appetite of the PWS patient is is controlled the method it will be able to prove the thing directly, it used the RIA kit and the ELISA it will be able to measure kit it will be able to measure the whole ghrelin to pick the PWS patient and the blood of the normal army and active ghrelin it measured a change.

DETAILED DESCRIPTION:
It will reach to respect, in 5 ' -flanking region of the ghrelin 2000 bp focus it let and it got luciferase assay it led and and it searched for the binding it sorted it put out and and to sleep the transcription factor which and and is the possibility of doing the essential region in the transcription and and it did an order deletion clone and and. is important in result and ghrelin activity the region role, -300~-200 region Basic helix-loop-helix (bHLH) are containing -USF (-236 to -231) binding site specially to be compressed in -500~-400 and -300~-200 two portions.

ELIGIBILITY:
Inclusion Criteria:

* PWS patients were genetically confirmed using the standard methylation test. GHD was diagnosed using a GH stimulation test. The lean and obese normal subjects (comparison group) enrolled were the children or siblings of hospital staff who understood the purpose of and the procedures used.

Exclusion Criteria:

* GHD patients had no history of GH treatment, and were not being treated with GH at study commencement

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Sixteen PWS patients [age, 8.1 +- 2.6 yr; 12 males, 4 females; body mass index (BMI), 25+-1.5 kg/m2], 19 healthy normal lean subjects (age, 8.9 +- 1.4 yr; 14 males, 5 females; BMI, 16.5 +- 0.42 kg/m2), 13 GHD patients (age, 9.1 +- 1.8 yr; 9 males, 4 females; BMI, 27 +- 1.8 kg/m2), and 10 healthy normal obese subjects (age, 8.7 +- 2.3 yr; 7 males, 3 females; BMI, 26 +- 1.7 kg/m2) were enrolled in the study. The subjects had no history of GH treatment and were not being treated with GH at study commencement.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2005-01; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Kyu Jin, M.D, Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine